CLINICAL TRIAL: NCT05843136
Title: Interferential Current Treatment Reduces Low Back Pain and Improves Functionality in Patients With Chronic Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Oeste do Para (Other)
Collaborators: Fundação Amazônia de Amparo a Estudos e Pesquisas FAPESPA (Unknown)
Responsible Party: Principal Investigator, LUIZ PAULO SOBRAL PEREIRA, Master's in Health Sciences, Universidade Federal do Oeste do Para
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAEE: 52035721.9.0000.0171
Record Dates: First submitted 2023-04-12; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Chronic Low-back Pain
Keywords: Interferential Current; Chronic low back pain; Quality of life; Occupational disease; Physical functionality
MeSH Terms: conditions — Occupational Diseases

STUDY DESIGN:
Intervention Model Description: The research is a randomized clinical trial, was submitted and approved by the Human Ethics Committee (CEP) with opinion 5,175,882, CAEE: 52035721.9.0000.0171. Participants were chosen at random, with single-blind masking, Random Allocation ® software was used to generate random numbers for the intervention and control groups, non-probalistic convenience sample. There were three groups: interventional, control 01 and control 02
Who Masked: Participant
Masking Description: only the participant was blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervenction (Experimental): We used the SONOPULSE II device from the manufacturer IBRAMED, the electrodes measuring nine centimeters in length and five centimeters in width, from the manufacturer ARKTUS, of the adhesive plate type.
  According to the IBRAMED manual (2011, p. 47), the application is produced by two medium frequency currents through four electrodes, quadripolar method. The current type is tetrapolar interferential and the stimulation mode is automatic vector; the carrier frequency of 4000HZ, AMF modulation frequency of 50HZ, and the sweep frequency of SWEEP will be 20HZ. SWEEP sweep modes with 6 seconds of rise from the modulation frequency to the threshold the sweep frequency upon reaching the threshold immediately decays over the next 6 seconds. The positioning of the four-leaf clover type electrodes and the intensity of the strong current, however comfortable, according to the patient's report.
  Interventions: Other: physiotherapy treatment
- Control Group 01 (Active Comparator): he treatment is based on non-invasive methods, highlighting manual therapy techniques, especially joint manipulation therapy. Manual therapy techniques are adjustments in lumbar rotation. Joint adjustment is a controlled lever-like force with direction, amplitude, and speed that is applied to specific, tissue-adjacent joints. While joint mobilization is manual therapy without the impulse, the joint remains within the physiological range of motion (SILVA et al., 2012). Therefore, a high-velocity, low-amplitude (HVA) manual maneuver was applied. The thrust (impulse) is carried out in the para-physiological environment, between the physiological and anatomical barriers. preload phase before the manipulation, thrust phase where the maneuver is performed with high speed and low amplitude and the resolution phase where the manipulation ends. The maneuver is detailed by the authors Bergmann & Peterson (2010).
  Interventions: Other: physiotherapy treatment
- Control Group 02 (Active Comparator): The procedure adopted in this group was based on the guidelines and recommendations for non-pharmacological treatment of the Associação Médica Brasileira AMB (RACHED, R.D.V.A. et al, 2013) use of 1 MHZ Ultrasound with a power of 1W/cm2, continuous IBRAMED device for 10 minutes, Wave Diathermy Short for 15 minutes/day, HTM brand, TENS 50 HZ and 50 ms intensity phase according to the patient's threshold, 30 minutes, IBRAMED brand
  Interventions: Other: physiotherapy treatment

INTERVENTIONS:
Other: physiotherapy treatment — this is an interventional study of the use of 3 physiotherapy treatment techniques in order to evaluate the effectiveness of interferential current in relieving chronic low back pain

SUMMARY:
. 24 individuals were evaluated, with low back pain for more than 12 weeks and aged between 12 and 65 years. The current used in the lumbar region of the participants was of the tetrapolar interferential type and the stimulation mode was the automatic vector, carrier of 4,000 HZ, modulation frequency (AMF) of 50 HZ, sweep frequency of SWEEP of 20HZ. The assessment of pain and functionality was performed using the data collection instrument, the Visual Analogue Pain Scale (VAS), Rolland Morris Disability Questionnaire (RMDQ) and the Owestry Disability Questionnaire (ODQ) respectively. The present study demonstrates that treatment with interferential current promotes chemical improvement in participants, which opens up new perspectives on the use of this therapeutic approach.

DETAILED DESCRIPTION:
Low back pain is characterized by pain and represents a change in health that affects mainly adults, although electrostimulation represents an important tool in the treatment of patients with chronic nonspecific low back pain, the clinical efficacy of the interferential current used in physiotherapy still lacks reinforcement for clinical validation. In this way, the present study evaluated whether the use of interferential current contributes to reducing chronic low back pain and analyzed whether the electrotherapeutic protocol can benefit the physical functionality of patients with chronic low back pain. 24 individuals were evaluated, with low back pain for more than 12 weeks and aged between 12 and 65 years. The current used in the lumbar region of the participants was of the tetrapolar interferential type and the stimulation mode was the automatic vector, carrier of 4,000 HZ, modulation frequency (AMF) of 50 HZ, sweep frequency of SWEEP of 20HZ. The assessment of pain and functionality was performed using the data collection instrument, the Visual Analogue Pain Scale (VAS), Rolland Morris Disability Questionnaire (RMDQ) and the Owestry Disability Questionnaire (ODQ) respectively. Data analysis was performed using the JAMOVI 2.2.5 software. Our data showed that individuals with interferential current showed significant improvement in pain relief, as well as in the functional pattern of pain improvement. The present study demonstrates that treatment with interferential current promotes chemical improvement in participants, which opens up new perspectives on the use of this therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both genders
* Aged between 18 and 65 years
* Voluntarily sought the Clinic's physiotherapy service
* Low back pain for more than 12 weeks
* Medical request and diagnosis of low back pain with or without pain radiating to the lower limbs
* Immunization against COVID 19.
* Signature of the free detailed term clarified. (FDTC)

Exclusion Criteria:

* Physiotherapy treatment carried out in a period equal to or less than 8 weeks before starting the research
* Reporting any contraindications inherent to the use of electrotherapy
* Participants with fractures or spinal surgery
* Involved in a legal medical dispute
* Diagnosis of fibromyalgia
* Patients with flu-like symptoms during the research period
* Participants who have more than 2 (two) absences will be excluded from the research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Isolated comparative evaluation method, before and after, in the three arms with Application of Rolland Morris Questionnaires | 12 months
  Application of Rolland Morris Questionnaires before and after intervention, this questionnaires assesses mild and moderate pain and disability
Isolated comparative evaluation method, before and after, in the three arms, Application of Owestry Questionnaire | 12 months
  Application of Owestry Questionnaire before and after intervention, this questionnaires evaluates more severe disabilities
Isolated comparative evaluation method, before and after, in the three arms, Application analogue visual score for pain | 12 months
  Application analogue visual score for pain before and after intervention, evaluates the level of pain according to the patient's reference

CONTACTS AND LOCATIONS:
Locations (1):
- Luiz Paulo Sobral Pereia, Santarém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: No